CLINICAL TRIAL: NCT01312168
Title: Endothelial Dysfunction, Monocyte Activation, and Vasculopathy in Patients With Obstructive Sleep Apnea and Effect of Six-month CPAP Treatment: A Large-scale, Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Endothelial Dysfunction, Monocyte Activation, and Vasculopathy in Patients With Obstructive Sleep Apnea (OSA) and Effect of 6-month CPAP Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: China Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201012085RB
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Sleep Apnea, Obstructive; Continuous Positive Airway Pressure; Endothelium; Inflammation; Vascular Function
Keywords: Cardiovascular disease; Continuous positive airway pressure; Endothelium; Vascular function; Inflammation; Sleep Apnea; Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive; Inflammation; Cardiovascular Diseases; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy non-OSA control (No Intervention)
- OSA receiving therapeutic CPAP (Experimental)
  Interventions: Device: Therapeutic CPAP
- OSA receiving subtherapeutic CPAP (Sham Comparator)
  Interventions: Device: Subtherapeutic CPAP

INTERVENTIONS:
Device: Therapeutic CPAP — CPAP ventilator, optimal pressure decided by CPAP manual titration, daily use at sleep, six months
  Arms: OSA receiving therapeutic CPAP
Device: Subtherapeutic CPAP — Subtherapeutic CPAP ventilator, pressure <3 cmH2O, daily use at sleep, six months
  Arms: OSA receiving subtherapeutic CPAP

SUMMARY:
This purpose of this study is to

1. Determine the change in endothelial dependent vascular reactivity and vascular properties
2. Determine the changes in monocytes activation
3. Determine the change in pro-inflammatory status
4. Investigate the effect of six-month CPAP therapy on the above changes in patients with OSA

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), characterized with chronic intermittent hypoxia (CIH) and sleep fragmentation, is associated with three-fold higher risk of cardiovascular events. CIH could promote production of ROS which induced the adhesion of circulating monocytes, endothelium injury, and production of pro-inflammatory mediators and adhesion molecules and lead to formation of atherosclerotic plaque. Recent studies showed vascular endothelium function could be noninvasively assessed with Flow-mediated dilation (FMD) in brachial artery, whereas OSA patients have lower FMD compared to control subjects. However, the CPAP effects on vascular function have conflicting results. Conflicts usually involve the small sample size, lack of appropriate control, and inadequate control of confounding factors, like physical activity, and duration of CPAP treatment. Also, CPAP effect on other monocytes activation and inflammatory mediators are clear as well. Our previous studies showed 12-week CPAP treatment could not modify the levels of TNF-α and hsCRP. However, the 12-week treatment may be not long enough to draw the conclusions for benefit from long-term CPAP therapy. Therefore, we plan to conduct a cross-sectional followed by a double blind, randomized, placebo-control, parallel-group interventional study to prove our hypothesis that OSA can lead to endothelial dysfunction, monocytes activation, and pro-inflammatory state which leads to and vasculopathy and those changes can be reverted by CPAP.

ELIGIBILITY:
OSA patients

Inclusion Criteria:

* male patients aged 30 to 65 year who have daytime sleepiness (ESS>=10)
* newly diagnosed OSA (AHI>30/hr) by overnight PSG but never been treated

Exclusion Criteria:

* unwilling or unable to perform testing procedure
* past or current smoking history
* medical condition (including cardiovascular disease, chronic pulmonary disease, diabetes, endocrinologic disease, chronic renal failure, and psychiatric disease)
* systemic inflammatory conditions (system lupus erythematosus, rheumatoid arthritis, sarcoidosis, Crohn's disease, and ulcerative colitis)
* active neurologic event
* active infection two weeks prior to screening
* enrolled in other trials in the study period
* other sleep disorders
* sleepy driver
* using maintenance medications

Control subjects

Inclusion Criteria:

* Age-, sex-, body weight-, height-matched subjects with enrolled OSA patients
* non-sleepy
* no OSA confirmed by home sleep study (AHI<5/hr)

Exclusion Criteria:

* unwilling or unable to perform testing procedure
* past or current smoking history
* medical condition (including cardiovascular disease, chronic pulmonary disease, diabetes, endocrinologic disease, chronic renal failure, and psychiatric disease)
* systemic inflammatory conditions (system lupus erythematosus, rheumatoid arthritis, sarcoidosis, Crohn's disease, and ulcerative colitis)
* active neurologic event
* active infection two weeks prior to screening
* enrolled in other trials in the study period
* other sleep disorders
* using maintenance medications

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2011-03; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
vascular reactivity of brachial artery and pulse wave velocity | six months

SECONDARY OUTCOMES:
percentage of adhesion molecule expression on monocytes | six months
levels of extra and intracellular cytokine | six months

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan